CLINICAL TRIAL: NCT02893085
Title: Tumor Mutation Profiling in Bile Samples From Patients With Biliary Strictures Related to Pancreatico-biliary Cancers
Brief Title: Pancreatico-biliary Tumor Mutation Profiling in Bile Samples
Acronym: ONCOBIL
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PA15117
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Cholangiocarcinoma, Cancer of the Head of the Pancreas
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Biomarkers; Vascular Endothelial Growth Factor A; Matrix Metalloproteinases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- patients with malignant biliary stricture
  Interventions: Biological: bile sample analysis; Biological: biochemical markers, VEGF and MMPs, in bile samples
- patients with benign biliary diseases
  Interventions: Biological: biochemical markers, VEGF and MMPs, in bile samples

INTERVENTIONS:
Biological: bile sample analysis — tumor mutation profile tumor genotype
  Groups: patients with malignant biliary stricture
Biological: biochemical markers, VEGF and MMPs, in bile samples

SUMMARY:
The differential diagnosis between benign and malignant bile duct strictures is a difficult and demanding task for clinicians. Clinical, biochemical, and radiological characteristics of malignant biliary strictures are non-specific and tissue diagnosis is difficult to obtain preoperatively. For this reason, there is a need for the development of new diagnostic modalities. Of particular interest is the quest of tumor markers secreted or shed in bile by tumor cells developing in the biliary tract.

In addition, patient's tumor molecular profile is the basis for selecting personalized therapy. Cholangiocarcinomas are characterized by a large genetic heterogeneity. The most frequent mutations are TP53, KRAS, BRAF, EGFR, MET, NRAS, PIK3CA, ERBB2, SMAD4, FBXW7, ARID1A, PBRM1, BAP1 et IDH1/2. In the case of pancreatic cancers, the most frequent are KRAS mutation detected in 90 % of the patients and CDKN2A, SMAD4, TGFBR1, TGFBR2, ATM, BRCA2, MLL2, MLL3, KDM6A, ARID1A, ARID1B, SMARC1, GNAS and RNF43 mutations.

It is well established that KRAS and P53 mutations can be detected in bile samples from patients with biliary strictures related to cholangiocarcinoma and cancer of the head of the pancreas. The main objective is to determine if bile sample analysis from patients with malignant biliary stricture may allow to identify tumor mutation profile and determine tumor genotype. A secondary objective is to evaluate the diagnostic value of Vascular Endothelial Growth Factor (VEGF) and metallo-proteinases (MMPs) levels in bile samples.

Tumor genotyping will be performed in bile samples (supernatant and cell pellet) and tumor tissues in a series of 10 patients surgically treated for malignant biliary stricture related to cholangiocarcinoma or cancer of the head of the pancreas. The biochemical markers, VEGF and MMPs, will be assessed in bile samples obtained during endoscopic retrograde cholangiopancreatography in 50 patients with malignant biliary stricture and 50 patients treated for benign biliary diseases.

ELIGIBILITY:
1. Tumor genotyping in bile samples:

   Inclusion criteria :
   * patients surgically treated for malignant biliary stricture related to cholangiocarcinoma or cancer of the head of the pancreas.
   * diagnosis of cholangiocarcinoma or cancer of the head of the pancreas confirmed by histopathological analysis of the resected specimen
   * adult patients

   Exclusion criteria :

   - patient who did not accept the storage of bile and tissue in the tissue Bank of Reims university hospital
2. Measurement of biochemical markers, VEGF and MMPs in bile samples obtained during endoscopic retrograde cholangiopancreatography in 50 patients with malignant biliary stricture and 50 patients treated for benign biliary diseases.

Inclusion criteria:

* patients with benign biliary diseases or malignant biliary stricture (cholangiocarcinoma or cancer of the head of the pancreas.
* indication of endoscopic retrograde cholangiopancreatography for diagnostic and therapeutic purposes
* adult patients Exclusion criteria
* patient who did not accept the storage of bile and tissue in the tissue Bank of Reims university hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with malignant biliary stricture and 50 patients with benign biliary diseases
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Tumor genotyping | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, France, Reims, France